CLINICAL TRIAL: NCT01142323
Title: Pilot Study of Fenofibrate in Primary Sclerosing Cholangitis
Brief Title: Pilot Study of Fenofibrate for PSC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: University of Florida (Other)
Responsible Party: Principal Investigator, Cynthia Levy, Associate Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20100533
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Results first posted 2013-04-23 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fenofibrate (Experimental): fenofibrate 160 mg po daily
  Interventions: Drug: fenofibrate

INTERVENTIONS:
Drug: fenofibrate — 160 mg po daily

SUMMARY:
The purpose of this study is to determine whether fenofibrate is safe and effective in the treatment primary sclerosing cholangitis (PSC).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of 18 to 75 years old
* Confirmed diagnosis of PSC including typical findings of stricturing and dilatations of the intra and/or extrahepatic biliary ducts in radiographic exam, (endoscopic retrograde cholangiopancreatography -ERCP, percutaneous cholangiogram - PTC or magnetic resonance cholangiopancreatography- MRCP)
* Serum alkaline phosphatase levels elevated to at least 1.5 times the upper limit of normal.

Exclusion Criteria:

* Hypersensitivity to fenofibrate
* Prisoners and institutionalized subjects
* Pregnant or nursing women
* Anticipated need for liver transplantation in one year
* Recipients of liver transplantation
* Recurrent variceal hemorrhage, uncontrolled encephalopathy or refractory ascites
* Co-existing liver diseases including auto-immune and viral hepatitis
* Acute or chronic renal failure, defined as glomerular filtration rate (GFR)< 60 ml/min, GFR calculated using the Modification of Diet in Renal Disease (MDRF) GFR calculator
* Known cholecystitis
* Current use of statins
* Current use of coumadin anticoagulant therapy
* Previous history of, or known high risk for, venous thromboembolism,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Levy, MD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fenofibrate
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fenofibrate
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Serum Alkaline Phosphatase
Description: Serum alkaline phosphatase will be measured at entry and end of study
Time Frame: 6 months
Measure: Median (Standard Error); unit: U/L
Groups:
- Baseline: Prior to drug intervention
- At 6 Months: fenofibrate 160 mg/day
Arm/Group | Baseline | At 6 Months
Number analyzed (Participants) | 8 | 8
U/L | 290 (76) | 165 (19)
Statistical Analysis 1: Comparison: Baseline vs At 6 Months; Test type: Superiority or Other; p = 0.008, Matched pairs

2. Secondary Outcome: Mayo Risk Score for Primary Sclerosing Cholangitis
Description: The Mayo risk score (MRS), which is a composite of several variables (age, bilirubin, albumin, aspartate aminotransferase[AST] and h/o variceal bleeding), will be measured at entry and end of study. The MRS is a mathematically calculated risk score.
  MRS does not have a theoretical lower/upper bound (that is, no theoretical minimum and maximum values).
  Mayo risk score <=0 indicates low risk of death. MRS between 0 and 2 indicates intermediate risk, and greater than 2 indicates high risk.
  There is no known range for this score.
Time Frame: 6 months
Population: Median baseline MRS was compared to Median MRS after 6 months of study drug
Measure: Median (Full Range); unit: score
Arm/Group | Fenofibrate
Number analyzed (Participants) | 8
score
  Baseline | -0.41 [-0.71 to 1.4]
  After 6 months | -0.46 [-0.96 to 1.8]
Statistical Analysis 1: Comparison: Fenofibrate; Test type: Superiority; p = 0.46, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Fenofibrate
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Fenofibrate (N=8)
worsening of psoriasis (Skin and subcutaneous tissue disorders) | 1/1 (1) — Only 1 patient had psoriasis at baseline, and therefore only 1 patient was at risk for worsening of Psoriasis. Of note, none of the other 7 patients developed new psoriasis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No